CLINICAL TRIAL: NCT01961284
Title: Zygomatic Versus Conventional Dental Implants in Augmented Maxillae: a Pragmatic Multicentre Randomised Clinical Trial.
Brief Title: Zygomatic Versus Conventional Dental Implants in Augmented Maxillae
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor company decision to terminate study
Sponsor: NHS Lothian (Other Government)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Victor Lopes, Professor Victor Lopes, Consultant in Oral and Maxillofacial surgery, NHS Lothian
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13/SS/0106
Record Dates: First submitted 2013-09-04; First posted 2013-10-11 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Edentulous Maxilla; Resorbed Maxilla; Implant Therapy

ARMS (2):
- Zygomatic Implants (Active Comparator): 2-4 zygomatic implants inserted into edentulous maxilla with no augmentation/grafting prior to providing patient with dental prosthesis
  Interventions: Device: Zygomatic implant placement
- Bone Graft and Conventional implants (Active Comparator): Edentulous maxilla which is deficient in bone is first grafted using bone grafting material derived from cows and then ordinary implants are placed into the augmented jaw bone approximately 6 monhts after grafting. Patients will be provided with a dental prosthesis following osseointegration.
  Interventions: Device: conventional implants and augmentation of maxilla

INTERVENTIONS:
Device: Zygomatic implant placement
  Arms: Zygomatic Implants
Device: conventional implants and augmentation of maxilla
  Arms: Bone Graft and Conventional implants

SUMMARY:
Dental implants are used for replacing missing teeth. Placing dental implants is limited by the presence of adequate bone volume permitting their anchorage. In order to solve this problem several bone augmentation procedures have been developed. In principle the missing bone is taken from a donor site (for example the hip), transplanted where needed and then implants are placed. Sometimes, major bone grafting operations have to be undertaken under general anaesthesia requiring patients to be hospitalised for a few days. Some degree of morbidity related to the donor site must be expected, though more recently bone substitutes are used to minimize morbidity, and 2 to 3 surgical interventions may be needed before the implants can be functionally used. Sometimes patients have to wait more than 1 year before a prosthesis can be fixed to the implants and the total cost of the treatment is high. At the beginning of the 1990s a long screwshaped implant was developed by Professor PI Brånemark as an alternative to bone augmentation procedures: the zygomatic implant. Zygomatic implants are generally inserted through the palate to engage the body of the cheek bone. One to three zygomatic implants can be inserted through the posterior palate to engage the body of each cheek bone. The potential main advantages of zygomatic implants could be that bone grafting may not be needed and a fixed prosthesis could be fitted the same day of their placement. Despite that zygomatic implants have been used for more than 20 years, their effectiveness has never been compared with conventional dental implants in augmented maxillae. The aim of the project is to compare the longtermclinical outcome of fullarch upper jaw bridges supported by zygomatic implants versus conventional implants placed in augmented bone in the palate.

ELIGIBILITY:
Inclusion Criteria:

* fully edentulous patients
* atrophic maxilla
* insufficient bone volume for placement of dental implants
* patients with no more than 4mm of bone height sub-antrally

Exclusion Criteria:

* general contraindications to implant surgery
* history of radiation therapy
* immunosuppressed/immunocompromised patients
* patients taking bisphosphonates
* poor oral hygiene
* patients with untreated periodontitis
* uncontrolled diabetes
* pregnancy
* alcohol/drug addiction
* lack of opposite occluding dentition/prosthesis
* restricted mouth opening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Implant success | 1 year following implant loading
  Implant failure is defined by implant mobility +/- infection dictating implant removal.
Implant success | 3 years following implant loading
  Implant failure is defined by implant mobility +/- infection dictating implant removal
Implant success | 5 years after implant loading
  Implant failure is defined by implant mobility +/- infection dictating implant removal.
Implant Success | 7 years after implant loading
  Implant failure is defined by implant mobility +/- infection dictating implant removal
Implant Success | 10 years after implant loading
  Implant failure is defined by implant mobility +/- infection dictating implant removal
Implant success | 15 years after implant loading
  Implant failure is defined by implant mobility +/- infection dictating implant removal

SECONDARY OUTCOMES:
Complications | 1 year
  Biologic and prosthetic complications will be assessed. Biologic complications include perimplantitis, maxillary sinusitis,abscess, fistula, gingival dehiscence.
  Prosthetic complication: abutment fracture
Change in marginal bone levels on intra oral radiographs | 1,3,5,7,10,15 years
  To be evaluated on intraoral radiographs taken with the paralleling technique at implant placement, at delivery of the provisional prostheses, 1, 3, 5, 7, 10 and 15 years after loading.
Failure of augmentation procedure | 6 months after augmentation procedure
  The augmentation procedure will be considered a failure if, after it has been performed, it will not be possible to place the planned implants in the augmented site.
Change in Oral Health impact profile OHIP-14 | 1,3,5,7,10,15
  To be filled in i)at patient enrolment prior to delivering any interventions, ii)12 weeks after delivery of the definitive prostheses and iii) 1, 3, 5, 7, 10 and 15 years after loading. Patients' number of days with total or partial impaired activity assessed at delivery of the provisional prosthesis A days of total impaired activity is one where patient is unable to perform his/her ordinary life activity including work. A days of partial impaired activity is one where the patient is only partially able to perform his/her ordinary life activity including work.
Complications | 3 years
  Biologic and prosthetic complications will be assessed. Biologic complications include perimplantitis, maxillary sinusitis, abscess, fistula, gingival dehiscence Prosthetic complication: abutment fracture
Complications | 5 years
  Biologic and prosthetic complications will be assessed. Biologic complications include perimplantitis, maxillary sinusitis, abscess, fistula, gingival dehiscence Prosthetic complication: abutment fracture
Complications | 7 years
  Biologic and prosthetic complications will be assessed. Biologic complications include perimplantitis, maxillary sinusitis, abscess, fistula, gingival dehiscence Prosthetic complication: abutment fracture
Complications | 10 years
  Biologic and prosthetic complications will be assessed. Biologic complications include perimplantitis, maxillary sinusitis, abscess, fistula, gingival dehiscence Prosthetic complication: abutment fracture
Complications | 15 years
  Biologic and prosthetic complications will be assessed. Biologic complications include perimplantitis, maxillary sinusitis, abscess, fistula, gingival dehiscence Prosthetic complication: abutment fracture

CONTACTS AND LOCATIONS:
Overall Officials: Victor Lopes, PhD, Study Chair — NHS Lothian
Locations (2):
- United Kingdom (2):
  - Glasgow Dental Hospital and School, Glasgow
  - St John's Hospital, Livingston